CLINICAL TRIAL: NCT06445270
Title: Evidence-informed Lifestyle Interventions to Improve Glycemic Parameters and Reduce Gestational Diabetes in High-risk Pregnant Individuals
Brief Title: Lifestyle Interventions to Improve Glycemic Parameters and Reduce Gestational Diabetes in High-risk Pregnant Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Northeastern University (Other); University of Texas (Other)
Responsible Party: Principal Investigator, David Haas, Munsick Professor of Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREVENT-GDM
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes; Pregnancy Complications
Keywords: gestational diabetes; prevention; pregnancy; continuous glucose monitor
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm consists of standard of care counseling for diet and exercise.
- GDM Prevention Program (Experimental): This arm consists of a more intensive exercise and monitoring program. .
  Interventions: Behavioral: GDM Prevention Program

INTERVENTIONS:
Behavioral: GDM Prevention Program — Participants will receive hybrid and group monthly contacts with registered dieticians and lifestyle coaches. Participants will attend monthly in-person physical activity sessions.
  Arms: GDM Prevention Program

SUMMARY:
The goal of this study is assess the impact of a higher intensity dietary and activity counseling program to improve blood sugar control and reduce the chance of developing gestational diabetes (GDM) as compared to the current standard diet and activity counseling.

DETAILED DESCRIPTION:
GDM is associated with adverse maternal and newborn outcomes, as well as potential lifelong consequences. Currently, clinical guidelines recommend screening for pre-existing Type 2 diabetes mellitus at new obstetric visits for individuals at high risk of developing GDM. For those who do not screen positive, but still may be at risk for GDM, standard practice is for basic diet, exercise, and weight gain counseling.

In this study, eligible participants will be randomized into one of two groups: usual care with standard diet and exercise counseling or a GDM prevention program that consists of a more intensive exercise and monitoring program.

All participants will be asked to wear an activity tracker and continuous glucose monitors (CGMs) at specified time points throughout their pregnancy. Blood will be drawn at specified time points to measure hemoglobin A1c, lipids, and HOMA-IR measures.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less or equal to 16 + 6 weeks confirmed via ACOG dating guidelines AND one of the following
* 35 years of age or older
* Family history of first degree relative with diabetes mellitus
* Body Mass Index (BMI) greater than or equal to 30
* Hemoglobin A1c value between 5.9% to 6.4%

Exclusion Criteria:

* Multiple gestations
* Current diagnosis of Type 1 or 2 diabetes mellitus including a diagnosis during this pregnancy
* Pre-pregnancy chronic (>2 weeks) usage of systemic steroids (inhaled and short term usage acceptable)
* Planned pregnancy termination
* Currently taking or took 3 months prior to conception Metformin
* Unable to provide informed consent in English or Spanish
* Major fetal anomalies listed below that are known prior to enrollment.

Major fetal anomalies:

* Congenital diaphragmatic hernia
* Congenital cystic adenomatoid malformation
* Pleural effustions
* Chylothorax
* Bronchogenic cyst
* Bronchopulmonary sequestration
* Anomalous pulmonary venous return
* Tricuspid atresia
* Mitral atresia
* Double right ventricle
* Ebstein's malformation
* Pulmonary atresia
* Hypoplastic left heart syndrome
* Aortic coarctation
* Fetal arrhythmias
* Transposition of the great vessels
* Tetrology of Fallot
* Double outlet right ventricle
* Aortic stenosis
* Holoprosencephaly
* Anencephaly
* Dandy-Walker malformation or variant
* Septo-optic dysplasia
* Neural tube defect
* Vein of Galen aneurysm
* Bilateral renal agenesis
* Cystic renal disease
* Obstructive uropathy
* Horseshoe kidney
* Megacystis microcolon
* Cloacal abnormality
* Achondrogenesis
* Thanatophoric dysplasia
* Thoracic dysplasia
* Osteogenesis imperfecta
* Short rib polydacyly
* Any skeletal defect with suspected small thorax
* Hypophosphatemia
* Any karyotypic abnormality
* Any suspected genetic syndrome
* Cleft lip/palate
* Micrognathia
* Hydrops
* Fetal anemia (<35% on cordocentesis)
* Neck mass
* Gastroschsis
* Omphalocele

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Time spent in euglycemia | 7 days per month
  percentage of time in a day spent in euglycemia

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No